CLINICAL TRIAL: NCT04870047
Title: Coating to Optimize Aneurysm Treatment In The New Flow Diverter Generation
Acronym: COATING
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Phenox GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO48/BO1309
Record Dates: First submitted 2021-04-26; First posted 2021-05-03 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- p64 MW HPC Flow Diverter + SAPT (Experimental)
  Interventions: Device: Endovascular treatment of unruptured aneurysms with p64 MW HPC Flow Modulation Device
- p64 MW Flow Diverter + DAPT (Experimental)
  Interventions: Device: Endovascular treatment of unruptured aneurysms with p64 MW HPC Flow Modulation Device

INTERVENTIONS:
Device: Endovascular treatment of unruptured aneurysms with p64 MW HPC Flow Modulation Device — Patients suffering from a distal intracranial aneurysm will be treated endovascularly with the p64 MW HPC Flow Modulation Device.

SUMMARY:
To assess safety and efficacy of p64 MW HPC Flow Modulation Device under single antiplatelet therapy compared to p64 MW Flow Modulation Device under dual antiplatelet therapy.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Subject has a saccular, unruptured or recanalized intracranial aneurysm. The subject may also have a previous ruptured aneurysm, provided rupture of this aneurysm 30 days from the index procedure.
3. Subject is intended to be treated for only one target aneurysm during the index procedure except for segmental disease (multiple aneurysms located on the same arterial segment aimed to be treated with one investigational device or investigational telescopic devices).
4. Subject has already been selected for flow diversion therapy as the appropriate treatment.
5. Subject has a mRS ≤ 2 before the procedure, as determined by a certified assessor independent of the index procedure.
6. Subject is able to understand the patient information and provides written informed consent verifying the use of his/her data (according to data protection laws).

Exclusion Criteria:

1. Subject who is currently prescribed under any long lasting antiplatelet and/or anticoagulation medication.
2. Subject has undergone a surgery including endovascular procedures in the last 30 days prior to the study procedure.
3. Subject has had an Intracranial hemorrhage and/or subarachnoid hemorrhage in the past 30 days prior to the study procedure.
4. Subject with target aneurysm previously treated with a stent or flow diverter.
5. Subject is expected to be treated for another aneurysm during the 30 days following the index procedure.
6. Subject with a confirmed stenosis in parent artery.
7. Subject with a blister-like aneurysm, fusiform aneurysm, dissecting aneurysm or aneurysm associated with a brain arteriovenous malformation (AVM).
8. Subject has a pre-procedure mRS >2.
9. Any known contraindication to treatment with the p64 MW HPC Flow Modulation Device in accordance with device IFU.
10. Subject who has undergone stenting of the ipsilateral carotid artery within 3 months of the index procedure.
11. Known serious sensitivity to radiographic contrast agents.
12. Known sensitivity to nickel, titanium metals, or their alloys.
13. Subject already enrolled in other clinical trials (including COATING study) that would interfere with study endpoints.
14. Known renal failure as defined by a serum creatinine > 2.5 mg/dl (or 220 μmol/l) or glomerular filtration rate (GFR) < 30.
15. Subject who has a contraindication to MRI or angiography for whatever reason.
16. Subject with a comorbid disease or condition that would confound the neurological and functional evaluations or compromise survival or ability to complete follow-up assessments.
17. Subject with any known allergy to heparin, ASA or other antiplatelet medications.
18. Subject with coagulation disorder
19. Pregnant woman or breast feeding.
20. Adults who lack the capacity to provide informed consent, and all those persons deprived of their liberty in prisons or other places of detention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of DWI lesions | 48 hours (± 24 hours)
  Number of diffusion-weighted imaging (DWI) lesions within 48 hours (+/- 24 hours) of the index procedure visualized via MRI.

SECONDARY OUTCOMES:
Short-term morbi-mortality rate | 30 days (± 7 days)
  Morbi-mortality rate at 30 days assessed by mRS > 2
Rate of neurological death or major stroke | 180 days (150 - 240 days) and 365 days (335 - 456 days) post procedure
  Rate of neurological death or major stroke (ischemic or hemorrhagic, defined as an increase of 4 or more points according to the National Institute of Health Stroke Scale Score) in the territory supplied by the treated artery, as assessed by the Clinical Events Committee
Long-term morbi-mortality rate | 180 days (150 - 240 days) and 365 days (335 - 456 days) post procedure
  Rate of subjects who have a mRS decline to a score of 3 or more (mRS > 3), or an increase of 2 points from baseline mRS score, as assessed by the Clinical Events Committee
Rate of subjects with dissusion-weighted imaging (DWI) lesions | 48 hours (± 24 hours)
  Rate of subjects with greater than 6 diffusion-weighted imaging (DWI) lesions or territorial stroke
Delayed aneurysm rupture | 180 days (150 - 240 days) and 365 days (335 - 456 days) post procedure
  Rate of an intracranial hemorrhage from delayed aneurysm rupture (from the day after index procedure), as assessed by the Clinical Events Committee
Delayed intraparenchymal hemorrhage | 180 days (150 - 240 days) and 365 days (335 - 456 days) post procedure
  Rate of delayed intraparenchymal haemorrhage unrelated to aneurysm rupture, as assessed by the Clinical Events Committee
Rate of peripheral bleeding | Any event reported from discharge to 365 days (335 - 456 days) post procedure
  Rate of peripheral bleeding, as assessed by the Clinical Events Committee
Rate of device deployment at the target site without technical complications | During intervention
  Rate of device deployment at the target site without technical complications, as assessed by the site
Rate of complete aneurysm occlusion | 180 days (150 - 240 days) and 365 days (335 - 456 days) post procedure
  Rate of complete aneurysm occlusion using the 3-grade scale, as assessed by the Core Lab
Rate of target aneurysm recurrence | 180 days (150 - 240 days) and 365 days (335 - 456 days) post procedure
  Rate of target aneurysm recurrence, as assessed by the Imaging Core Lab
Rate of target aneurysm retreatment | 180 days (150 - 240 days) and 365 days (335 - 456 days) post procedure
  Rate of target aneurysm retreatment, as assessed by the Clinical Event Committee
Rate of intrastent stenosis and/or thrombosis at the target site | 180 days (150 - 240 days) and 365 days (335 - 456 days) post procedure
  Rate of intrastent stenosis and/or thrombosis at the target site, as assessed by the Core Lab through DSA
Mean length of hospital stay | From admission up to discharge, assessed up to 456 days
  Mean length of hospital stay (from hospital admission and up to hospital discharge)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Pierot, Prof. Dr., Principal Investigator — CHRU Hôpital Maison-Blanche
Locations (18):
- France (5):
  - CHU Bordeaux, Bordeaux
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHU de Lyon, Lyon
  - CHU de Montpellier, Montpellier
  - CHU Reims - Hôpital Maison Blanche, Reims
- Germany (7):
  - Universitätsklinikum Augsburg, Augsburg
  - Helios Klinikum Erfurt, Erfurt
  - Universitätsklinikum Halle (Saale), Halle
  - Klinikum der LMU München, München
  - Klinikum Nürnberg Süd, Nuremberg
  - Klinikum Vest Recklinghausen, Recklinghausen
  - Klinikum Stuttgart, Stuttgart
- Hadassah University Medical Center, Jerusalem, Israel
- Fondazione I.R.C.C.S. Instituto Neurologico Carlo Besta, Milan, Italy
- UNLP Košice, Košice, Slovakia
- Universitätsspital Basel, Basel, Switzerland
- United Kingdom (2):
  - Queen Elisabeth Hospital Birmingham, Birmingham
  - Western General Hospital, Edinburgh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramirez-Velandia F, Enriquez-Marulanda A, Filo J, Young M, Fodor TB, Sconzo D, Muram S, Granstein JH, Shutran M, Taussky P, Ogilvy CS. Comparison of Thromboembolic Events Between Pipeline Embolization Device (PED) Shield and PED/PED Flex: A Propensity Score-Matched Analysis. Neurosurgery. 2024 Aug 1;95(2):330-338. doi: 10.1227/neu.0000000000002883. Epub 2024 Feb 23. PMID 38391195
- [Derived] Pierot L, Lamin S, Barreau X, Berlis A, Ciceri E, Cohen JE, Costalat V, Eker OF, Henkes H, Holtmannspotter M, Januel AC, Keston P, Klisch J, Psychogios MN, Valvassori L, Cognard C, Spelle L. Coating (Coating to Optimize Aneurysm Treatment in the New Flow Diverter Generation) study. The first randomized controlled trial evaluating a coated flow diverter (p64 MW HPC): study design. J Neurointerv Surg. 2023 Jul;15(7):684-688. doi: 10.1136/neurintsurg-2022-018969. Epub 2022 May 24. PMID 35609974